CLINICAL TRIAL: NCT06326853
Title: Neuroendocrine Mechanisms in Adiposity: An Integrated Approach to the Characterization of Potential Pharmacological Novel Targets Based on Experimental and Clinical Models
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Giustina, Professor of Endocrinology and Metabolism, IRCCS San Raffaele
Other Study IDs: Adipofisi
Record Dates: First submitted 2024-03-18; First posted 2024-03-22 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Endocrine Disorders; Adiposity; Pituitary Adenoma; Cushing Syndrome; Acromegaly; Hypopituitarism
MeSH Terms: conditions — Endocrine System Diseases; Obesity; Pituitary Neoplasms; Cushing Syndrome; Acromegaly; Hypopituitarism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients affected by hypothalamic-pituitary endocrine pathology: 100 patients affected by hypothalamic-pituitary endocrine pathology who have performed or who will perform a first visit at the Endocrinology Department of the San Raffaele Hospital between 01/01/2021 and 31/12/2026.
- affected by obesity: 100 patients affected by obesity who will perform a first visit at the Endocrinology Department of the San Raffaele Hospital between 01/01/2021 and 31/12/2026.

SUMMARY:
The goal of this observational study is to evaluate, retrospectively and prospectively, the effect of different hormonal and neuropeptide dysfunctions on the body composition of patients suffering from hypothalamic-pituitary pathologies, and to evaluate the potential beneficial effect of surgical and medical treatments with agonists and antagonists of hypothalamic neuropeptides, currently available, on the development and treatment of adiposity and negative cross-talk between adiposity and muscle/bone tissue

ELIGIBILITY:
Inclusion Criteria:

Obese patients affected and not by hypothalamic-pituitary diseases

Exclusion Criteria:

1. Minor subjects;
2. Pregnant and/or breastfeeding women;
3. Patients suffering from states of primary and/or acquired immunodeficiencies, and/or serious impairment of general clinical conditions (e.g. metastatic neoplasms; immunosuppressive therapies; worsening/reacerbated/compensated chronic pathologies);
4. Patients unable to understand and sign the Informed Consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by: Non-secreting pituitary adenomas, Prolactinoma, Cushing's disease, Acromegaly, TSHomas, hypopituirarisms treated with cabergoline, octreotide, lanreotide, pasireotide, pegvisomant, rhGH and/or undergoing surgical therapy (transnasosphenoidal neurosurgical removal of the pituitary tumor. Healthy obese subjects.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with BMI greater than 30 with hypothalamic-pituitary pathologies | retrospective and prospective collection of clinical data between 01/01/2021 and 31/12/2026
  The study aims to evaluate, retrospectively and prospectively, the effect of different hormonal and neuropeptide dysfunctions on the body composition of patients suffering from hypothalamic-pituitary pathologies